CLINICAL TRIAL: NCT02774694
Title: Observational Study of the Nociceptive Flexion Reflex Threshold to Predict Outcome After Interventional Pain Management Procedures in Patients With Chronic Back and Neck Pain. A Study of Diagnostic Accuracy
Brief Title: Prediction of Outcome of Interventional Pain Management
Acronym: POINTPM
Status: Not yet recruiting | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, Médecin adjoint agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 15-072
Record Dates: First submitted 2015-12-02; First posted 2016-05-17 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Neck Pain; Chronic Pain
Keywords: nociceptive flexion reflex; interventional pain management
MeSH Terms: conditions — Low Back Pain; Neck Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational cohort: patients undergoing interventional pain management procedures
  Interventions: Device: nociceptive flexion reflex (NFR) threshold ("Paintracker", Dolosys GmbH, Berlin, Germany)

INTERVENTIONS:
Device: nociceptive flexion reflex (NFR) threshold ("Paintracker", Dolosys GmbH, Berlin, Germany) — measurement of the NFR threshold using the "Paintracker" device
  Other Names: R3 reflex

SUMMARY:
Interventional pain management for back and neck pain is widely used, but the indications and relative merits of these techniques rest subject to discussion. This study aims to identify prognostic criteria for patients who might specifically benefit from interventional pain management. Specifically, the nociceptive reflex threshold will be investigated, which is a measure of central sensibilisation and thus a potentially important prognostic factor.

DETAILED DESCRIPTION:
Interventional pain management is resource-intensive and carries non-negligible risks. Not all patients profit equally from such procedures. For those who do not benefit, the risk of potential complications is futile, and the resources are wasted. Therefore, a possibility to distinguish responding patients from non-responders would be important.

Central pain sensitization has been related to poor outcome, and electrical pain and reflex thresholds are a good measure of pain hypersensitivity at least in chronic low back pain. Especially the nociceptive flexion reflex (NFR) threshold has been identified to correlate well with central pain hypersensibility. Successful interventional pain treatment has been shown to reverse central hypersensibility as measured by the NFR threshold.

NFR threshold, in contrast to pain threshold, seems to be a measure independent of psychological factors. Thus the NFR threshold could give information independent of psychological factors in order to predict poor outcome of interventional pain management procedures.

The study will be a prospective observational trial of diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic low back or neck pain (duration >3 months)
* scheduled for the following interventions: epidural injection, facet block, medial branch block, facet radiofrequency denervation, spinal cord stimulator implantation

Exclusion Criteria:

* inability to understand the patient information or the study questionnaires
* patients <18 years old
* patients with implanted pacemakers or defibrillators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included will be patients treated by the interventional pain management team of the department of anaesthesiology of the Geneva University Hospitals HUG
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
ROC-AUC for incidence of pain reduction>30% at 1 week | 1 week
  Primary study outcome is the diagnostic accuracy of the NFR threshold, measured as area under the "receiver operating characteristic ROC" curve, for the following main pain management outcome:
  "pain reduction of 30% one week after the interventional procedure

SECONDARY OUTCOMES:
ROC-AUC for incidence of pain reduction>30% at 1 month | 1 month
  Area Under the curve (AUC) of the receiver-operating characteristic (ROC) of the relation between NFR reflex threshold and the incidence of pain reduction>30% at 1 month
ROC-AUC for incidence of pain reduction>30% at 3 months | 3 months
  Area Under the curve (AUC) of the receiver-operating characteristic (ROC) of the relation between NFR reflex threshold and the incidence of pain reduction>30% at 3 months
ROC-AUC for incidence of pain reduction>30% at 6 months | 6 months
  Area Under the curve (AUC) of the receiver-operating characteristic (ROC) of the relation between NFR reflex threshold and the incidence of pain reduction>30% at 6 months
ROC-AUC for physical functioning at 1 week | 1 week
ROC-AUC for emotional functioning at 1 week | 1 week
ROC-AUC for patient rating of improvement and satisfaction at 1 week | 1 week
adverse events of interventional pain management | 1 week
patient disposition at 1 week, 1,3, and 6 months | 6 months
  The presence or unexcused absence of the patient at each consultation visit is noted

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: Undecided